CLINICAL TRIAL: NCT00668564
Title: Treatment of Lysosomal and Peroxisomal Inborn Errors of Metabolism by Hematopoietic Cell Transplantation
Brief Title: Hematopoietic Stem Cell Transplantation (HCT) for Inborn Errors of Metabolism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by another study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2008-02; 0801M25202 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hurler's Syndrome; Maroteaux-Lamy Syndrome; Sly Syndrome; Alpha Mannosidosis; Fucosidosis; Aspartylglucosaminuria; Sphingolipidoses; Krabbe Disease; Wolman's Disease; Niemann-Pick Disease Type B; Niemann-Pick Disease, Type C
Keywords: Inborn errors of metabolism; Sphingolipidoses; Recessive Leukodystrophies- GLD, Krabbe disease, MLD; Peroxisomal Disorders; Wolman syndrome; Niemann-Pick B patients; Niemann-Pick C subtype 2
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; alpha-Mannosidosis; Fucosidosis; Aspartylglucosaminuria; Sphingolipidoses; Leukodystrophy, Globoid Cell; Wolman Disease; Niemann-Pick Disease, Type B; Niemann-Pick Disease, Type C; Metabolism, Inborn Errors; Leukodystrophy, Metachromatic; Peroxisomal Disorders | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Cyclophosphamide; Alemtuzumab; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intent-to-Treat (Experimental): All patients treated with study regimen.
  Interventions: Procedure: Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Campath-1H; Drug: Busulfan

INTERVENTIONS:
Procedure: Stem Cell Transplantation — The purpose of hematopoietic stem cell transplantation is to introduce blood producing cells from a normal donor. These cells can either provide what is missing in the body to the other cells, or can change the body's immune response to the substances that have accumulated in the body. These normal hematopoietic stem cells can come from bone marrow, peripheral blood (i.e., the blood circulating in our body's blood vessels) or umbilical cord blood (i.e., blood taken from the umbilical cord after a baby is born and umbilical cord is cut). The new donor cells repopulate the blood and bone marrow system and enter the organs of the body, including the brain. Wherever these cells go, they will produce the needed enzyme.
  Other Names: Bone Marrow Transplant, cord blood transplant
Drug: Cyclophosphamide — Days before Transplant Drug Frequency
  * 4 Cyclophosphamide Once, given over 2 hours
  * 3 Cyclophosphamide Once, given over 2 hours
  * 2 Cyclophosphamide Once, given over 2 hours
  * 1 Cyclophosphamide Once, given over 2 hours
  Other Names: Cytoxan
Drug: Campath-1H — Days before Transplant Drug Frequency
  12 Campath-1H Once, given over 2 hours
  11 Campath-1H Once, given over 2 hours
  10 Campath-1H Once, given over 2 hours
  Other Names: Alemtuzamab
Drug: Busulfan — Days before Transplant Drug Frequency
  9 Busulfan Four times per day
  8 Busulfan Four times per day
  7 Busulfan Four times per day
  6 Busulfan Four times per day
  Other Names: Busulfex

SUMMARY:
The primary objective of this clinical trial is to evaluate the ability to achieve and sustain donor engraftment in patients with lysosomal and peroxisomal inborn errors of metabolism undergoing hematopoietic stem cell transplantation (HCT).

DETAILED DESCRIPTION:
This has been an ongoing area of interest by our group at the Univ. of Minnesota, but this is a new protocol to take the place of several older protocols. While survival has been very good on the prior protocols over the past decade, incomplete engraftment has remained somewhat problematic. Therefore, we have modified the preparative regimen somewhat to increase engraftment by replacing anti-thymocyte globulin (ATG) with Campath-1H, a drug that is more immune suppressive. In addition, we have modified the supportive care regimen. Based on this, we will monitor levels of an anti-oxidant therapy (N-acetylcysteine) and biomarkers of inflammation and oxidative stress for the families that consent to these research studies.

ELIGIBILITY:
Inclusion Criteria:

* Mucopolysaccharidosis (MPS) Disorders:

  * MPS IH (Hurler syndrome)
  * MPS-VI (Maroteaux-Lamy syndrome)
  * MPS VII (Sly syndrome).
* Glycoprotein metabolic disorders:

  * Alpha mannosidosis
  * Fucosidosis
  * Aspartylglucosaminuria
* Sphingolipidoses and Recessive Leukodystrophies: Presymptomatic patients with globoid cell leukodystrophy (GLD, also known as Krabbe disease) and metachromatic leukodystrophy (MLD) will be eligible for treatment on this protocol. White matter disease by magnetic resonance imaging (MRI) alone is not an exclusion if the patient is asymptomatic.
* Peroxisomal Disorders: Presymptomatic patients with inherited peroxisomal disorders associated with of very long chain fatty acids (VLCFA) elevation, identified by family history or laboratory testing (including neonatal screening), are eligible for this protocol. White matter disease by MRI alone is not an exclusion if the patient is asymptomatic.
* Other Inherited Diseases of Metabolism:

  * Wolman syndrome (acid lipase deficiency)
  * Niemann-Pick B patients (sphingomyelin deficiency)
  * Niemann-Pick C subtype 2
* Donor Availability: Patients considered for transplantation must have a sufficient graft as based on current criteria of the University of Minnesota Blood and Marrow Transplantation Program: Priority will be as follows, although in circumstances in which timing is of the essence, cord blood grafts may be chosen over an unrelated graft, despite the priority listed above.
* Multidisciplinary Evaluation: Patients will be eligible for transplantation only after they are seen and evaluated by members of the Inherited Metabolic and Storage Disease Program (IMSD) team, and the team has offered transplantation to the patient/family.

Exclusion Criteria:

* Symptomatic patients with peroxisomal or lysosomal disorders are excluded but may be considered for other treatment protocols.
* Major organ dysfunction. Evidence of major organ impairment, including:

  * Cardiac: left ventricular ejection fraction <40%
  * Renal: serum creatinine >2.5 x normal for age
  * Hepatic: total bilirubin >3 x normal, or Alanine transaminase (ALT) > 3 x normal
  * Pulmonary: requirement for continuous oxygen supplementation
* Pregnancy
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* Patients >21 years of age.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — University of Minnesota Medical Center
Locations (1):
- University of Minnesota, Fairview, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miller WP, Rothman SM, Nascene D, Kivisto T, DeFor TE, Ziegler RS, Eisengart J, Leiser K, Raymond G, Lund TC, Tolar J, Orchard PJ. Outcomes after allogeneic hematopoietic cell transplantation for childhood cerebral adrenoleukodystrophy: the largest single-institution cohort report. Blood. 2011 Aug 18;118(7):1971-8. doi: 10.1182/blood-2011-01-329235. Epub 2011 May 17. PMID 21586746

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent-to-Treat: All patients treated with study regimen; Bone Marrow Transplant - cord blood transplant; Cyclophosphamide (50 mg/kg intravenous [IV] days 1-4 prior to transplant); Busulfan (if < or = 12 kg: 1.1 mg/kg or if > 12 kg: 0.8 mg/kg IV every 6 hours on days 6-9 before transplant) and Campath-1H (once per day 0.3 mg/kg IV on days 10-12 before transplant.
Period: Overall Study
Arm/Group | Intent-to-Treat
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Engraftment
Description: Rate of successful engraftment - patients who achieved and sustained donor engraftment; donor chimerism by day 100 of at least 90% after undergoing hematopoietic stem cell transplantation.
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 18
Participants | 14

2. Secondary Outcome: Overall Survival
Description: Number of patients alive at timepoints.
Time Frame: Day 100, 1 Year, 3 Years
Population: Year 3 survival endpoint was not done due to study being terminated prematurely.
Measure: Number; unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 18
Participants
  Day 100 | 14
  1 Year | 12

ADVERSE EVENTS:
Time Frame: Day 1 through Day 100 post-transplant.
Description: Only Serious Adverse Events were collected for this study.
Arm/Group | Intent-to-Treat
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=18)
Death (General disorders) | 6 (6)
Graft failure (Blood and lymphatic system disorders) | 2 (2)
Auto recovery (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Other secondary objectives outlined in study protocol were not analyzed; number of patients were too few to be relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes